CLINICAL TRIAL: NCT05089188
Title: PRAME Immunohistochemistry as an Adjunct for Evaluating Ambiguous Melanocytic Proliferation
Acronym: ANTIPRAME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8420
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Melanoma
Keywords: Immunohistochemistry; Histopathology
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunomarkers — immunohistochemical expression profile of ambiguous melanocytic proliferation.

SUMMARY:
Skin melanoma is a common form of skin cancer. Its diagnosis is usually clinically suspected and then affirmed by histopathological examination.

In some cases, the histopathological analysis of these lesions is equivocal, and the malignant or benign nature of the proliferation is difficult to determine with certainty. In these cases, the use of expensive ancillary tests, which are hardly accessible and take a long time to set up (FISH - CGH-array), is usually required.

Anti-PRAME immunostaining, an inexpensive and readily available technic, has recently been described as highly sensitive and specific for diagnosing malignant melanocytic proliferations. Knowledge on its utility for evaluating ambiguous melanocytic neoplasms remains limited.

Our study aims to improve the current body of knowledge on the utility of PRAME immunohistochemistry for evaluating challenging samples of melanocytic proliferation. The secondary objective is to determine the PRAME immunoreactivity profile for each histological subtype of melanocytic proliferations (spitzoid tumors, cellular blue nevi, dysplastic nevi ...)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient at the time of diagnosis (> = 18 years).
* histopathological diagnosis of "ambiguous melanocytic proliferation" or "atypical melanocytic proliferation" made between January 2016 and December 2020.
* Histological slides archived in the "CRB" biobank available
* Formalin-fixed paraffin-embedded tissue block archived in the "CRB" biobank available
* Informed patient

Exclusion Criteria:

* Patient who has expressed opposition to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases with histopathological diagnosis of "ambiguous melanocytic proliferation" or "atypical melanocytic proliferation" made between January 2016 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Immunomarkers | 1 month
  Correlation of melanocytic lesions' histopathological diagnosis concerning benignity or malignancy with anti-PRAME immunohistochemical expression profile

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided